CLINICAL TRIAL: NCT00998868
Title: Observational Study to Evaluate the Prevalence of Rotator Cuff Tears in Hemiplegic Shoulders
Brief Title: Rotator Cuff Tears in Hemiplegic Shoulder
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Other Study IDs: SNUH-RM-TRHan-RCTHS-01
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Hemiplegia
Keywords: Rotator Cuff; Tendinopathy; ultrasonography
MeSH Terms: conditions — Hemiplegia; Tendinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hemiplegia: patients with hemiplegia, without other musculoskeletal disorders of the shoulder

SUMMARY:
The purpose of the study is to evaluate the prevalence of rotator cuff tears in the shoulders of hemiplegic patients of different severity.

DETAILED DESCRIPTION:
Rotator cuff tears are often suspected to contribute hemiplegic shoulder pain. However, it is controversial whether their incidence increases in hemiplegia. Based on the postulate that muscle weakness in hemiplegia predisposes rotator cuff injury due to biomechanical failure, this study aims to investigate whether the rotator cuff tears are associated with the muscle strength of the shoulder by observing hemiplegic shoulders of varying degree of paresis.

ELIGIBILITY:
Inclusion Criteria:

* hemiplegia; unilateral weakness of sudden onset
* secondary to strokes or other brain lesions
* compatible with brain lesions confirmed by imaging studies

Exclusion Criteria:

* bilateral weakness
* any history of intensive trauma of the shoulder, reported
* preexisting musculoskeletal disorder of the shoulder

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: university hospital, department of rehabilitation medicine admitted patients due to hemiplegia
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tai Ryoon Han, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Reilly P, Macleod I, Macfarlane R, Windley J, Emery RJ. Dead men and radiologists don't lie: a review of cadaveric and radiological studies of rotator cuff tear prevalence. Ann R Coll Surg Engl. 2006 Mar;88(2):116-21. doi: 10.1308/003588406X94968. PMID 16551396
- [Background] Sano H, Ishii H, Trudel G, Uhthoff HK. Histologic evidence of degeneration at the insertion of 3 rotator cuff tendons: a comparative study with human cadaveric shoulders. J Shoulder Elbow Surg. 1999 Nov-Dec;8(6):574-9. doi: 10.1016/s1058-2746(99)90092-7. PMID 10633891
- [Background] Yu D. Shoulder pain in hemiplegia. Phys Med Rehabil Clin N Am. 2004 Aug;15(3):vi-vii, 683-97. doi: 10.1016/S1047-9651(03)00130-X. PMID 15219895
- [Background] Bender L, McKenna K. Hemiplegic shoulder pain: defining the problem and its management. Disabil Rehabil. 2001 Nov 10;23(16):698-705. doi: 10.1080/09638280110062149. PMID 11732559
- [Background] Gilmore PE, Spaulding SJ, Vandervoort AA. Hemiplegic shoulder pain: implications for occupational therapy treatment. Can J Occup Ther. 2004 Feb;71(1):36-46. doi: 10.1177/000841740407100108. PMID 15015899
- [Background] Van Ouwenaller C, Laplace PM, Chantraine A. Painful shoulder in hemiplegia. Arch Phys Med Rehabil. 1986 Jan;67(1):23-6. PMID 3942479
- [Background] Joynt RL. The source of shoulder pain in hemiplegia. Arch Phys Med Rehabil. 1992 May;73(5):409-13. PMID 1580765
- [Background] Hakuno A, Sashika H, Ohkawa T, Itoh R. Arthrographic findings in hemiplegic shoulders. Arch Phys Med Rehabil. 1984 Nov;65(11):706-11. PMID 6497618
- [Background] Rizk TE, Christopher RP, Pinals RS, Salazar JE, Higgins C. Arthrographic studies in painful hemiplegic shoulders. Arch Phys Med Rehabil. 1984 May;65(5):254-6. PMID 6712451
- [Background] Lo SF, Chen SY, Lin HC, Jim YF, Meng NH, Kao MJ. Arthrographic and clinical findings in patients with hemiplegic shoulder pain. Arch Phys Med Rehabil. 2003 Dec;84(12):1786-91. doi: 10.1016/s0003-9993(03)00408-8. PMID 14669184
- [Background] Najenson T, Yacubovich E, Pikielni SS. Rotator cuff injury in shoulder joints of hemiplegic patients. Scand J Rehabil Med. 1971;3(3):131-7. No abstract available. PMID 5156175
- [Background] Nepomuceno CS, Miller JM 3rd. Shoulder arthrography in hemiplegic patients. Arch Phys Med Rehabil. 1974 Feb;55(2):49-51. No abstract available. PMID 4810651
- [Background] Wolff AB, Sethi P, Sutton KM, Covey AS, Magit DP, Medvecky M. Partial-thickness rotator cuff tears. J Am Acad Orthop Surg. 2006 Dec;14(13):715-25. doi: 10.5435/00124635-200612000-00003. PMID 17148619
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder. 1972. J Bone Joint Surg Am. 2005 Jun;87(6):1399. doi: 10.2106/JBJS.8706.cl. PMID 15930554
- [Background] MacGillivray JD, Fealy S, Potter HG, O'Brien SJ. Multiplanar analysis of acromion morphology. Am J Sports Med. 1998 Nov-Dec;26(6):836-40. doi: 10.1177/03635465980260061701. PMID 9850788
- [Background] Wang JC, Horner G, Brown ED, Shapiro MS. The relationship between acromial morphology and conservative treatment of patients with impingement syndrome. Orthopedics. 2000 Jun;23(6):557-9. doi: 10.3928/0147-7447-20000601-12. PMID 10875415
- [Background] Neer CS 2nd. Impingement lesions. Clin Orthop Relat Res. 1983 Mar;(173):70-7. No abstract available. PMID 6825348
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890
- [Background] Jobe CM. Superior glenoid impingement. Orthop Clin North Am. 1997 Apr;28(2):137-43. doi: 10.1016/s0030-5898(05)70274-1. PMID 9113710
- [Background] Blevins FT. Rotator cuff pathology in athletes. Sports Med. 1997 Sep;24(3):205-20. doi: 10.2165/00007256-199724030-00009. PMID 9327536
- [Background] Soslowsky LJ, Thomopoulos S, Tun S, Flanagan CL, Keefer CC, Mastaw J, Carpenter JE. Neer Award 1999. Overuse activity injures the supraspinatus tendon in an animal model: a histologic and biomechanical study. J Shoulder Elbow Surg. 2000 Mar-Apr;9(2):79-84. PMID 10810684
- [Background] Perry SM, McIlhenny SE, Hoffman MC, Soslowsky LJ. Inflammatory and angiogenic mRNA levels are altered in a supraspinatus tendon overuse animal model. J Shoulder Elbow Surg. 2005 Jan-Feb;14(1 Suppl S):79S-83S. doi: 10.1016/j.jse.2004.09.020. PMID 15726091
- [Background] Lohr JF, Uhthoff HK. The microvascular pattern of the supraspinatus tendon. Clin Orthop Relat Res. 1990 May;(254):35-8. PMID 2323147
- [Background] Rothman RH, Parke WW. The vascular anatomy of the rotator cuff. Clin Orthop Relat Res. 1965 Jul-Aug;41:176-86. No abstract available. PMID 5832730
- [Background] Rathbun JB, Macnab I. The microvascular pattern of the rotator cuff. J Bone Joint Surg Br. 1970 Aug;52(3):540-53. No abstract available. PMID 5455089
- [Background] Yuan J, Murrell GA, Wei AQ, Wang MX. Apoptosis in rotator cuff tendonopathy. J Orthop Res. 2002 Nov;20(6):1372-9. doi: 10.1016/S0736-0266(02)00075-X. PMID 12472255
- [Background] Yuan J, Murrell GA, Trickett A, Wang MX. Involvement of cytochrome c release and caspase-3 activation in the oxidative stress-induced apoptosis in human tendon fibroblasts. Biochim Biophys Acta. 2003 Jun 17;1641(1):35-41. doi: 10.1016/s0167-4889(03)00047-8. PMID 12788227
- [Background] Yuan J, Murrell GA, Trickett A, Landtmeters M, Knoops B, Wang MX. Overexpression of antioxidant enzyme peroxiredoxin 5 protects human tendon cells against apoptosis and loss of cellular function during oxidative stress. Biochim Biophys Acta. 2004 Jul 23;1693(1):37-45. doi: 10.1016/j.bbamcr.2004.04.006. PMID 15276323
- [Background] Bonita R, Beaglehole R. Recovery of motor function after stroke. Stroke. 1988 Dec;19(12):1497-500. doi: 10.1161/01.str.19.12.1497. PMID 3201508
- [Background] Soslowsky LJ, Malicky DM, Blasier RB. Active and passive factors in inferior glenohumeral stabilization: a biomechanical model. J Shoulder Elbow Surg. 1997 Jul-Aug;6(4):371-9. doi: 10.1016/s1058-2746(97)90005-7. PMID 9285877
- [Background] Ovesen J, Nielsen S. Experimental distal subluxation in the glenohumeral joint. Arch Orthop Trauma Surg (1978). 1985;104(2):78-81. doi: 10.1007/BF00454241. PMID 4051701
- [Background] Halder AM, Halder CG, Zhao KD, O'Driscoll SW, Morrey BF, An KN. Dynamic inferior stabilizers of the shoulder joint. Clin Biomech (Bristol). 2001 Feb;16(2):138-43. doi: 10.1016/s0268-0033(00)00077-2. PMID 11222932
- [Background] Niessen M, Janssen T, Meskers C, Koppe P, Konijnenbelt M, Veeger D. Kinematics of the contralateral and ipsilateral shoulder: a possible relationship with post-stroke shoulder pain. J Rehabil Med. 2008 Jun;40(6):482-6. doi: 10.2340/16501977-0201. PMID 18509565
- [Background] Diederichsen LP, Norregaard J, Dyhre-Poulsen P, Winther A, Tufekovic G, Bandholm T, Rasmussen LR, Krogsgaard M. The activity pattern of shoulder muscles in subjects with and without subacromial impingement. J Electromyogr Kinesiol. 2009 Oct;19(5):789-99. doi: 10.1016/j.jelekin.2008.08.006. Epub 2008 Dec 4. PMID 19062307
- [Background] Gold GE, Pappas GP, Blemker SS, Whalen ST, Campbell G, McAdams TA, Beaulieu CF. Abduction and external rotation in shoulder impingement: an open MR study on healthy volunteers initial experience. Radiology. 2007 Sep;244(3):815-22. doi: 10.1148/radiol.2443060998. Epub 2007 Aug 9. PMID 17690321
- [Background] Pong YP, Wang LY, Wang L, Leong CP, Huang YC, Chen YK. Sonography of the shoulder in hemiplegic patients undergoing rehabilitation after a recent stroke. J Clin Ultrasound. 2009 May;37(4):199-205. doi: 10.1002/jcu.20573. PMID 19253350
- [Background] Kim HA, Kim SH, Seo YI. Ultrasonographic findings of painful shoulders and correlation between physical examination and ultrasonographic rotator cuff tear. Mod Rheumatol. 2007;17(3):213-9. doi: 10.1007/s10165-007-0577-8. Epub 2007 Jun 20. PMID 17564776

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Jan, 2008 - Dec, 2009 Recruitment site: Seoul National University Eligible canditates from: inpatients in the department of rehabilitation medicine of the hospital Methods of recruitment: research physicians informed about the study to all eligible candidates and asked if they agreed to participate.
Pre-assignment Details: The study was designed to recruit hemiplegic patients of diverse degree of paresis with the same size. Because the crude distribution of the motor weakness was not even, the recruitment process adjusted the distribution of the severity of paresis, by recruiting patients of different motor strength in a consecutive way.
Period: Overall Study
Arm/Group | Hemiplegia
Started | 51 (>=10 for each muscle strength per MRC scale, after excluding the cases following exclusion criteria)
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hemiplegia
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 63.37 (10.765)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 25
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 51

OUTCOME MEASURES:

1. Primary Outcome: Rotator Cuff Tear of the Hemiplegic Shoulder, Confirmed by Ultrasonography
Description: All patients underwent ultrasonography (USG) for the both, affected and unaffected, shoulders. USG routinely examined biceps, subscapularis, supraspinatus, and infraspinatus tendons as for the partial or complete tears, calcifications, bony irregularity and bursal swellings.
Time Frame: within one month after enrollment
Measure: Number; unit: participants
Arm/Group | Hemiplegia
Number analyzed (Participants) | 51
participants | 29

2. Secondary Outcome: Rotator Cuff Tear of the Unaffected Shoulder, Confirmed by Ultrasonography
Description: All patients were performed ultrasonography (USG) for the both, affected and unaffected, shoulders. USG routinely examined biceps, subscapularis, supraspinatus, and infraspinatus tendons as for the partial or complete tears, calcifications, bony irregularity and bursal swellings.
Time Frame: within one month after enrollment
Measure: Number; unit: participants
Arm/Group | Hemiplegia
Number analyzed (Participants) | 51
participants | 18

3. Secondary Outcome: Subluxation of the Glenohumeral Joint, Confirmed by Physical Examination
Description: The glenohumeral joint subluxation was examined by palpating the subacromial regions of the both sides and comparing the affected side with the unaffected side while patients are seated and relaxed. If the palpated space between the acromion and the humeral head was wider on the affected side by one half finger breath or more, it was judged to be subluxation.
Time Frame: within one month after enrollment
Measure: Number; unit: participants
Arm/Group | Hemiplegia
Number analyzed (Participants) | 51
participants | 21

4. Secondary Outcome: Muscle Strength, Measured by Physical Examination, Per Medical Research Council Muscle Strength Grading System
Description: Muscle strength was measured for forward flexion and abduction of the shoulder per Medical Research Council (MRC) scale in each participants. Their mean +/- SD were calculated in each group.
  MRC scale:
  Grade 5: Normal and can move against full resistance. Grade 4: Reduced but can move against resistance. Grade 3: Can move only against gravity Grade 2: Can move without gravity Grade 1: Only a trace of movement Grade 0: No movement.
Time Frame: within one month after enrollment
Measure: Mean (Standard Deviation); unit: Units on a scale (minimum 0, maximum 5)
Arm/Group | Hemiplegia
Number analyzed (Participants) | 51
Units on a scale (minimum 0, maximum 5) | 1.96 (1.442)

ADVERSE EVENTS:
Arm/Group | Hemiplegia
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No